CLINICAL TRIAL: NCT02754739
Title: Effect of Pravastatin in the Subjects With Prediabetes or Early Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Collaborators: Daiichi Sankyo Korea Co., Ltd. (Industry)
Responsible Party: Principal Investigator, MOON-KYU LEE, M.D., Ph.D., Samsung Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2012-12-103
Record Dates: First submitted 2016-04-09; First posted 2016-04-28 (Estimated); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: Diabetes Mellitus; Prediabetic State
Keywords: Pravastatin; Insulin Resistance
MeSH Terms: conditions — Diabetes Mellitus; Prediabetic State; Insulin Resistance | interventions — Pravastatin

STUDY DESIGN:
Masking Description: This study was initially designed as a single center, double-blind, placebo-controlled, 2-group factorial randomized trial (placebo or pravastatin 40mg once daily for 24 weeks). Subjects were randomly assigned, in a 1:1 ratio, to receive pravastatin in a blinded fashion at a dose of 40 mg once daily or placebo. However, because of the problem of expiration date of the placebo drug, the study was converted to an open-label trial, and subjects without any medications were enrolled in an open-label control group in contrast to the pravastatin group. Therefore, the study cohort comprised the pravastatin group, placebo group, and the open-label control group. The placebo group and the open-label control group were classified as the control group.
Oversight: Data Monitoring Committee: No

ARMS (3):
- Pravastatin (Experimental): Pravastatin 40mg tablet by mouth, once daily for 24 weeks. Also, nutritional education was provided to participants in all arms by a nutritionist, and participants were instructed to follow the educated guideline.
  Interventions: Drug: Pravastatin
- Placebo (Placebo Comparator): Placebo drug indistiguishable from pravastatin 40mg tablet, by mouth, once daily for 24 weeks. Also, nutritional education was provided to participants in all arms by a nutritionist, and participants were instructed to follow the educated guideline.
  Interventions: Drug: Placebo (for Pravastatin)
- Open-label control (Other): No medication. Only nutritional education was provided to participants by a nutritionist, and participants were instructed to follow the educated guideline.
  Interventions: Behavioral: Nutritional education only

INTERVENTIONS:
Drug: Pravastatin — Pravastatin 40mg once daily for 24 weeks and nutritional education by a nutritionist
  Arms: Pravastatin
Drug: Placebo (for Pravastatin) — Pill manufactured to mimic pravastatin 40mg tablet once daily for 24 weeks and nutritional education by a nutritionist
  Arms: Placebo
Behavioral: Nutritional education only — Only nutritional education by a nutritionist
  Other Names: Open-label control
  Arms: Open-label control

SUMMARY:
An increased risk of incident diabetes with statin therapy have been reported in several studies. However, it is not recommended to limit the use of statin for this reason since the absolute risk increase was small, and the cardiovascular event rate reduction with statins overweighed the risk of new diabetes (Scatter N et al. Lancet, 2010). Moreover, each statin may have different effect on the development of incident diabetes. In the West of Scotland Coronary Prevention Study, pravastatin therapy reduced the hazard of becoming diabetic by 30%. Also, with pravastatin use, an increase in adiponectin level, which is related to the improvement in insulin sensitivity, has been reported. In this clinical trial, the investigators are aiming to evaluate the effect of pravastatin on insulin resistance, insulin secretion, glycemic control, and adiponectin level in participants with prediabetes or early diabetes by assigning them in a 24 weeks of pravastatin therapy group or in a placebo group.

ELIGIBILITY:
Inclusion Criteria:

* Subjects have early diabetes mellitus or prediabetes. Early diabetes mellitus or prediabetes are defined according to the following criteria; Subjects have two or more of the following three, or they have one of them at the initial test and the repeat test.

  1. hemoglobin A1C 5.7-9.0%
  2. fasting plasma glucose level 100mg/dL or more
  3. plasma glucose level 140mg/dL or more at 2 hours after 75g oral glucose tolerance test
* Subjects have one of the following three;

  1. Low-density lipoprotein cholesterol (LDL-cholesterol) 130mg/dL or more, and body mass index (BMI) > 23 kg/m2,
  2. 10 year atherosclerotic cardiovascular disease (ASCVD) risk of 7.5% or more, which is assessed by the ASCVD-Risk-Estimator (Circulation.2014;129:S1-S45)
  3. In diabetic patients, LDL-cholesterol 100mg/dL or more

Exclusion Criteria:

* Hemoglobin A1C > 9.0%
* History of statin use in three months
* Use of oral antidiabetic drugs except for metformin in three months
* History of malignant diseases (cancers)
* History of coronary artery diseases, heart failure, arrhythmia, valvular heart diseases, or cerebrovascular diseases
* Pregnant
* serum creatinine level > 1.5 mg/dL
* aspartate aminotransferase (AST) or alanine aminotransferase (ALT) levels higher than 80 U/l
* Taking weight loss medications, corticosteroids, Angiotensin converting enzyme (ACE) inhibitors, or estrogen replacement therapy
* Chronic hepatitis B or chronic hepatitis C

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2014-04-15 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
Insulin resistance assessed by HOMA-IR (homeostatic model assessment index for insulin resistance) | at the end of the 24 weeks of medication period
  compared to the HOMA-IR level calculated at the initial visit (at the beginning of the 24 weeks of medication period)

SECONDARY OUTCOMES:
Insulin resistance assessed by Matsuda index calculated through 75g oral glucose tolerance test | at the end of the 24 weeks of medication period
  calculated according to a method described in a previous study (Matsuda M et al. Diabetes Care, 1999), compared to the results at the initial visit (at the beginning of the 24 weeks of medication period). It takes 120 minutes to perform 75g oral glucose tolerance test
Insulin secretion capacity assessed by insulinogenic index (INS index) during 75g oral glucose tolerance test | at the end of the 24 weeks of medication period
  the ratio relating enhancement of circulating insulin in 30min [in pmol/L] to magnitude of corresponding glycemic stimulus in 30min [in mmol/L] during the oral glucose tolerance test (H.S. Seltze et al. J. Clin. Investig., 1967), compared to the results at the initial visit (at the beginning of the 24 weeks of medication period)
Insulin resistance assessed by the quantitative insulin sensitivity check index (QUICKI) | at the end of the 24 weeks of medication period
  calculated using fasting insulin in uIU/mL and fasting plasma glucose in mg/dL according to the method described in a previous study (A. Katz et al. J. Clin. Endocrinol. Metab., 2000), compared to the results at the initial visit (at the beginning of the 24 weeks of medication period)
Insulin secretory capacity relative to insulin resistance assessed by the oral disposition index | at the end of the 24 weeks of medication period
  calculated according to a method described in a previous study (K.M. Utzschneider et al.Diabetes Care, 2008), compared to the results at the initial visit (at the beginning of the 24 weeks of medication period)
Glycemic control evaluated by fasting glucose level (mg/dL) | at the end of the 24 weeks of medication period
  compared to the values at the initial visit
Glycemic control evaluated by hemoglobin A1C (%) | at the end of the 24 weeks of medication period
  compared to the values at the initial visit
Plasma adioponectin level (μg/ml), an adipocyte-derived insulin-sensitizing hormone level | at the end of the 24 weeks of medication period
  compared to the values at the initial visit
Biomarkers predicting cardiovascular diseases, assessed by high sensitive C-reactive protein (hsCRP) (mg/dL) | at the end of the 24 weeks of medication period
  compared to the values at the initial visit
Biomarkers predicting cardiovascular diseases, assessed by plasminogen activator inhibitor-1 (PAI-1) (ng/mL) | at the end of the 24 weeks of medication period
  compared to the values at the initial visit

CONTACTS AND LOCATIONS:
Overall Officials: Moon-Kyu Lee, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Division of Endocrinology and Metabolism, Department of Internal Medicine, Samsung Medical Center, Sungkyunkwan University School of Medicine, Seoul, South Korea

REFERENCES:
- [Background] Sattar N, Preiss D, Murray HM, Welsh P, Buckley BM, de Craen AJ, Seshasai SR, McMurray JJ, Freeman DJ, Jukema JW, Macfarlane PW, Packard CJ, Stott DJ, Westendorp RG, Shepherd J, Davis BR, Pressel SL, Marchioli R, Marfisi RM, Maggioni AP, Tavazzi L, Tognoni G, Kjekshus J, Pedersen TR, Cook TJ, Gotto AM, Clearfield MB, Downs JR, Nakamura H, Ohashi Y, Mizuno K, Ray KK, Ford I. Statins and risk of incident diabetes: a collaborative meta-analysis of randomised statin trials. Lancet. 2010 Feb 27;375(9716):735-42. doi: 10.1016/S0140-6736(09)61965-6. Epub 2010 Feb 16. PMID 20167359
- [Background] Rajpathak SN, Kumbhani DJ, Crandall J, Barzilai N, Alderman M, Ridker PM. Statin therapy and risk of developing type 2 diabetes: a meta-analysis. Diabetes Care. 2009 Oct;32(10):1924-9. doi: 10.2337/dc09-0738. PMID 19794004
- [Background] Freeman DJ, Norrie J, Sattar N, Neely RD, Cobbe SM, Ford I, Isles C, Lorimer AR, Macfarlane PW, McKillop JH, Packard CJ, Shepherd J, Gaw A. Pravastatin and the development of diabetes mellitus: evidence for a protective treatment effect in the West of Scotland Coronary Prevention Study. Circulation. 2001 Jan 23;103(3):357-62. doi: 10.1161/01.cir.103.3.357. PMID 11157685
- [Background] Guclu F, Ozmen B, Hekimsoy Z, Kirmaz C. Effects of a statin group drug, pravastatin, on the insulin resistance in patients with metabolic syndrome. Biomed Pharmacother. 2004 Dec;58(10):614-8. doi: 10.1016/j.biopha.2004.09.005. PMID 15589072
- [Background] Matsuda M, DeFronzo RA. Insulin sensitivity indices obtained from oral glucose tolerance testing: comparison with the euglycemic insulin clamp. Diabetes Care. 1999 Sep;22(9):1462-70. doi: 10.2337/diacare.22.9.1462. PMID 10480510
- [Background] Seltzer HS, Allen EW, Herron AL Jr, Brennan MT. Insulin secretion in response to glycemic stimulus: relation of delayed initial release to carbohydrate intolerance in mild diabetes mellitus. J Clin Invest. 1967 Mar;46(3):323-35. doi: 10.1172/JCI105534. PMID 6023769
- [Background] Katz A, Nambi SS, Mather K, Baron AD, Follmann DA, Sullivan G, Quon MJ. Quantitative insulin sensitivity check index: a simple, accurate method for assessing insulin sensitivity in humans. J Clin Endocrinol Metab. 2000 Jul;85(7):2402-10. doi: 10.1210/jcem.85.7.6661. PMID 10902785
- [Background] Utzschneider KM, Prigeon RL, Faulenbach MV, Tong J, Carr DB, Boyko EJ, Leonetti DL, McNeely MJ, Fujimoto WY, Kahn SE. Oral disposition index predicts the development of future diabetes above and beyond fasting and 2-h glucose levels. Diabetes Care. 2009 Feb;32(2):335-41. doi: 10.2337/dc08-1478. Epub 2008 Oct 28. PMID 18957530